CLINICAL TRIAL: NCT01275105
Title: A Single-Center, Randomized, Double-Masked, Placebo and Active Controlled, Dose-Ranging Evaluation of the Duration of Action of Brimonidine Tartrate Ophthalmic Solution in the Control of Ocular Redness Induced by Conjunctival Allergen Challenge (CAC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eye Therapies, LLC (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-100-0008
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vehicle (Other)
  Interventions: Drug: Vehicle
- Brimonidine Tartrate 0.01% (Active Comparator)
  Interventions: Drug: Brimonidine Tartrate 0.01%
- Oxymetazoline HCl 0.025% (Active Comparator)
  Interventions: Drug: Oxymetazoline HCl 0.025%
- Brimonidine Tartrate 0.025% (Active Comparator)
  Interventions: Drug: Brimonidine Tartrate 0.025%

INTERVENTIONS:
Drug: Vehicle — one drop in each eye at designated visits
  Arms: Vehicle
Drug: Brimonidine Tartrate 0.01% — one drop in each eye at designated visits
  Arms: Brimonidine Tartrate 0.01%
Drug: Brimonidine Tartrate 0.025% — one drop in each eye at designated visits
  Arms: Brimonidine Tartrate 0.025%
Drug: Oxymetazoline HCl 0.025% — one drop in each eye at designated visits
  Arms: Oxymetazoline HCl 0.025%

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and dose response of brimonidine tartrate ophthalmic solution as compared to placebo in the prevention of allergen-induced conjunctival redness using a conjunctival allergen challenge (CAC) model.

It is hypothesized that low-dose brimonidine tartrate ophthalmic solution will be more effective than vehicle in the prevention of conjunctival redness induced by conjunctival allergen challenge when instilled prior to the allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* If female, cannot be not pregnant or nursing
* Have a positive skin test reaction to cat hair, cat dander, grasses, ragweed, dog dander, cockroach, dust mite, and/or trees within the past 24 months;
* Have a calculated best corrected visual acuity of 0.6 logMAR or better in each eye as measured using an ETDRS chart;

Exclusion Criteria:

* Have known contraindications or sensitivities to the use of any of the study medications(s) or their components;
* Have any ocular condition that, in the opinion of the investigator, could affect the subject's safety;
* Have a presence of active ocular infection;
* Use specified disallowed medications during the study or appropriate pre-study washout period;
* Have any significant illness;
* Have planned surgery (ocular or systemic) during the trial period or within 30 days after;
* Have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device study within 30 days of the study;
* Be a female who is currently pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Conjunctival Redness | at specified timepoints for up to 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ora, Inc., Andover, Massachusetts, United States